CLINICAL TRIAL: NCT05200715
Title: Development of an International Multicenter Registry of Patients With Monogenic and Polygenic Autoinflammatory Diseases Aimed at Clinical and Therapeutical Data Collection and Analysis
Brief Title: AutoInflammatory Disease Alliance Registry (AIDA)
Acronym: AIDA
Status: Recruiting | Type: Observational
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Luca Cantarini, MD, PhD, Professor of Rheumatology, University of Siena
Other Study IDs: AIDA V.04 19.05.2021
Record Dates: First submitted 2021-12-18; First posted 2022-01-21 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Hereditary Autoinflammatory Diseases; Schnitzler Syndrome; Behcet Syndrome; PFAPA Syndrome; Still Disease; Autoinflammatory Syndrome, Unspecified; Uveitis; Scleritis; Vexas Syndrome; Spondyloarthritis (SpA); Castleman Disease
MeSH Terms: conditions — Hereditary Autoinflammatory Diseases; Schnitzler Syndrome; Behcet Syndrome; Marshall syndrome; Arthritis, Juvenile; Uveitis; Scleritis; VEXAS syndrome; Spondylarthritis; Castleman Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Patients affected by autoinflammatory diseases
  Interventions: Other: No intervention is foreseen by the protocol.

INTERVENTIONS:
Other: No intervention is foreseen by the protocol. — Patients will be observed for 10 years at least. Demographic, genetic, clinical, clinimetric, laboratory, radiologic and therapeutic data will be collected both retrospectively and prospectively during routine follow-up visits.

SUMMARY:
Autoinflammatory diseases (AID) are clinical entities characterized by recurrent inflammatory attacks in absence of infection, neoplasm or deregulation of the adaptive immune system. Among them, hereditary periodic syndromes, also known as monogenic AID, represent the prototype of this disease group, caused by mutations in genes involved in the regulation of innate immunity, inflammation and cell death. Based on recent experimental acquisitions in the field of monogenic AID, several immunologic disorders have been reclassified as polygenic/multifactorial AID, sharing pathogenetic and clinical features with hereditary periodic fevers. This has paved the way to new treatment targets for patients suffering from rare diseases of unknown origin, including Behçet's disease, Still disease, Schnitzler's disease, PFAPA (periodic fever, aphthous stomatitis, pharyngitis and cervical adenitis) syndrome, chronic recurrent multifocal osteomyelitis (CRMO), non-infectious uveitis and scleritis. Gathering information on such rare conditions is made difficult by the small number of patients, along with the difficulty of obtaining an accurate diagnosis in non-specialized clinical settings.

In this context, the AIDA project promotes international collaboration among clinical centres to develop a permanent registry aimed at collecting demographic, genetic, clinical and therapeutic data of patients affected by monogenic and polygenic AID, in order to expand the current knowledge of these rare conditions.

DETAILED DESCRIPTION:
The AIDA registry service is based on REDCap (Research Electronic Data Capture, project-redcap.org), a secure web application for building and managing online surveys and databases, designed to support data capture for research studies. The platform is directly accessible through the AIDA website, after inserting a personal username and password. Currently, 11 registries are available, each one dedicated to the collection of data about:

* monogenic AID
* PFAPA syndrome
* undifferentiated systemic AID (USAID)
* Behçet's disease
* Schnitzler's disease
* VEXAS (vacuoles, E1 enzyme, X-linked, autoinflammatory, somatic) syndrome
* Still disease
* noninfectious uveitis
* noninfectious scleritis
* spondyloarthritis
* Castleman disease

The registry will pursue the following aims within the first 36 months from the start of the enrollment:

1. to identify any association between clinical manifestations and gender, disease duration, body mass index and tabagism;
2. to detect differences in the clinical phenotype between pediatric-onset and adult-onset patients;
3. to identify the impact of different treatment approaches on clinical and laboratory disease manifestations.

Additional aims of the AIDA project, to be reached over the next 10 years, are the following:

1. to overcome fragmentation in the clinical experience on these rare conditions by sharing the knowledge at the international level;
2. to improve knowledge about the clinical presentation, genotype-phenotype correlations, response to treatment, long-term complications and social impact when monogenic and polygenic AID manifest during either childhood or adulthood;
3. to identify the long-term clinical course of patients diagnosed with monogenic or polygenic AID;
4. to promote awareness among physicians and enhance early recognition of these diseases;
5. to describe the impact of AID on quality of life;
6. to identify any impact of monogenic and polygenic AID on fertility;
7. to study the course of AID during pregnancy;
8. to assess the socioeconomic impact of AID;
9. to promote future multicentric studies.

Data collection is both retrospective and prospective. It includes demographic, clinical, diagnostic, genetic, clinimetric, laboratory, radiologic, therapeutic and socio-economic data. Instruments are designed to be filled out during routine clinical visits, usually scheduled every 3-6 months. Separation of personally identifiable information and medical data by using only pseudonyms for storing medical data ensures compliance with data protection regulations. The description of symptoms, diseases, procedures and injuries is based on the International Statistical Classification of Diseases and Related Health Problems (ICD)-10 coding system. Data management is both central and decentral. Data are extracted and statistically analyzed on a regular basis according to individual study protocols. A policy for authorship and dissemination of research findings is in place among the AIDA partners contributing to the registry.

The AIDA registry will support data collection for the conduction of clinical trials, observational studies, comparative effectiveness research, and other research on patients with monogenic and polygenic AID.

Several healthcare providers contributing to the AIDA Network are members of the European Reference Network (ERN) for Rare Immunodeficiency, Autoinflammatory and Autoimmune Diseases (RITA).

ELIGIBILITY:
Inclusion Criteria:

* to be diagnosed with a monogenic AID according to the clinical phenotype and the detection of a confirmative genotype;
* to be diagnosed with clinical familial Mediterranean fever or Behçet's disease or Still disease or PFAPA syndrome or Schnitzler's disease or CRMO according to the corresponding clinical diagnostic and/or classification criteria;
* to be diagnosed with undifferentiated systemic AID;
* to be diagnosed with non-infectious uveitis according to the standardization for uveitis nomenclature (SUN) criteria;
* to be diagnosed with anterior or posterior non-infectious scleritis;
* to be diagnosed with spondyloarthritis according to ASAS and/or New York criteria;
* to be diagnosed with Castleman disease;

Exclusion Criteria:

- informed consent/assent not provided by the patient and/or his/her legal representative.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients consecutively diagnosed and treated at the hospitals/ research centres affiliated to the AIDA Network (https://aidanetwork.org/en/)
Sampling Method: Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2020-08-06 (Actual); Primary Completion 2026-08-06 (Estimated); Study Completion 2030-08-06 (Estimated)

PRIMARY OUTCOMES:
Change of the number of enrolled subjects | 0-36-60-120 months
  This is an observational registry. The primary outcome is the increase of the number of subjects enrolled within each nosologic group.

SECONDARY OUTCOMES:
Change in the disease activity score | 0-36-60-120 months
  Change in the disease activity score specific for the nosologic entity (BDCAF score, Pouchot score, modified Pouchot score, JADAS27/JADAS27(CRP), DAS28) or according to composite indexes that will be defined in each study based on the registry.
Change in the % of patients with new organ involvement | 0-36-60-120 months
Incidence of death or adverse events | 0-36-60-120 months
Change in the inflammatory markers values (ESR) | 0-36-60-120 months
  ESR measured in mm/h
Change in the inflammatory markers values (CRP and SAA) | 0-36-60-120
  CRP and SAA measured in mg/dl
Change in visual acuity expressed as Best Corrected Visual Acuity (BCVA) | 0-36-60-120 months
Change in the overall function score | 0-36-60-120 months
  Change in the overall function score according to HAQ (adults) or CHAQ (children)
Change in the overall damage score | 0-36-60-120 months
  Change in the overall damage score specific for the nosologic entity (ADDI score, BODI score, JADI score)
Change in articular pain measured as Visual Analogue Scale for articular Pain (VAS Pain) | 0-36-60-120 months
Changes in height and weight percentile values for age and sex | 0-36-60-120 months
Change in the % of patients experiencing fatigue | 0-36-60-120 months
Change in the % of patients with fertility reduction or pregnancy complications | 0-36-60-120
Change in the socioeconomic indicators | 0-36-60-120 months
  Number of days lost at work/school during the last 3 months, Number of visits/ phone calls to the general practitioner during the last 3 months, Number of accesses to the Emergency Room during the last 6 months, Days of hospitalization during the last 3 months, Overall number of days lost at work by relatives during the last 3 months

CONTACTS AND LOCATIONS:
Locations (108):
- Algeria (2):
  - University Algiers 1, Algiers
  - Université M'Hamed Bougara de Boumerdas, Boumerdas
- Australia (2):
  - Flinders University, Adelaide
  - University of Adelaide, Adelaide
- Antwerp University Hospital, Antwerp, Belgium
- Hospital das Clinicas da Faculdade de Medicina HCFMUSP, São Paulo, Brazil
- China (2):
  - Peking University People's Hospital, Beijing
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
- Universidad del Rosario - Escuela de Medicina Y Ciencias de La Salud, Bogotá, Colombia
- Egypt (3):
  - Mansoura University, Faculty of Medicine, Al Mansurah
  - Al-Azhar University, Cairo
  - Cairo University, Cairo
- Universitätsklinikum Schleswig-Holstein, Lübeck, Germany
- Greece (2):
  - Evangelismos General Hospital, Athens
  - National and Kapodistrian University of Athens, Athens
- India (2):
  - Prabha Eye Clinic & Research Centre, Bangalore
  - Postgraduate Institute of Medical Education and Research, Chandigarh
- Shariati Hospital - Tehran University of Medical Sciences, Tehran, Iran
- Italy (59):
  - Azienda Ospedaliero-Universitaria Senese, Siena, Tuscany
  - AOUC Policlinico di Bari, Bari
  - University of Bari Medical School, Bari
  - University-Hospital of Bari - UOC Medicina Interna, Bari
  - University-Hospital of Bari - UOC Pediatria, Bari
  - University-Hospital of Bari - UOC Reumatologia, Bari
  - Central Hospital of Bolzano, Bolzano
  - ASST degli Spedali Civili - P.O. Ospedale dei Bambini, Brescia
  - ASST degli Spedali Civili, Brescia
  - Azienda Ospedaliera Universitaria di Cagliari, Cagliari
  - AOU Policlinico Vittorio Emanuele - Dip. Materno-Infantile, Catania
  - ARNAS Garibaldi - Catania, Catania
  - Azienda Ospedaliera di Catanzaro Pugliese Ciaccio, Catanzaro
  - Ospedale SS Annunziata, Chieti
  - Ospedale San Paolo, Civitavecchia
  - Arcispedale Sant'Anna, Ferrara
  - Azienda Ospedaliera Universitaria Careggi - SOD Medicina Interna Interdisciplinare, Florence
  - Azienda Ospedaliero-Universitaria Careggi - SOD Immunologia e Terapie Cellulari, Florence
  - Azienda Ospedaliero-Universitaria Meyer, Florence
  - Azienza Ospedaliero-Universitaria Careggi - SOD Reumatologia, Florence
  - Ospedale San Giovanni di Dio, Florence
  - Sapienza University - Polo Pontino, Latina
  - Ospedale Vito Fazzi, Lecce
  - ASL1 Avezzano, Sulmona, L'Aquila, L’Aquila
  - Università degli Studi di L'Aquila - UOC Medicina Interna e Nefrologia, L’Aquila
  - AOU Policlinico G. Martino, Messina
  - ASST Gaetano Pini/ CTO, Milan
  - Policlinico di Milano, Milan
  - ASST Fatebenefratelli Sacco - UO Medicina Generale, Milan
  - ASST Fatebenefratelli Sacco - UOC Reumatologia, Milan
  - ASST Gaetano Pini/CTO, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Ospedale Fatebenefratelli e Oftalmico, Milan
  - AORN Cardarelli, Napoli
  - AOU Federico II, Napoli
  - AOU Luigi Vanvitelli - UO Reumatologia, Napoli
  - AOU Luigi Vanvitelli - UOC Pediatria 2, Napoli
  - Azienda Ospedaliera Universitaria di Padova, Padua
  - ARNAS Civico Di Cristina Benfratelli, Palermo
  - ARNAS Ospedale Civico di Cristina Benfratelli, Palermo
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia-Cervello, Palermo
  - Università degli Studi di Palermo, Palermo
  - Fondazione IRRCS San Matteo - SC Reumatologia, Pavia
  - Azienda Ospedaliera di Perugia, Perugia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - University of Pisa, Pisa
  - AOU Policlinico Umberto I, Roma
  - Azienda Ospedaliera San Camillo Forlanini, Roma
  - IRCCS Fondazione PU Agostino Gemelli - UOC Medicina Interna Columbus, Roma
  - IRCCS Fondazione PU Agostino Gemelli - UOC Pediatria, Roma
  - Ospedale Pediatrico Bambino Gesù, Roma
  - Ospedale Universitario Campus Bio-Medico, Roma
  - Sapienza University - Polo Pontino, Roma
  - Università di Roma Tor Vergata, Roma
  - Azienda Ospedaliera Universitaria di Salerno, Salerno
  - ATS Sardegna, Tempio Pausania
  - AO Ordine Mauriziano, Torino
  - A.S.L. Vercelli - Ospedale S. Andrea, Vercelli
  - Azienda Ospedaliera Universitaria Integrata, Verona
- Tripoli Children Hospital, Tripoli, Libya
- University Hospital of Martinique, Fort-de-France, Martinique
- Mexico (2):
  - Asociacion para Evitar la Ceguera en México, Mexico City
  - Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City
- Poland (2):
  - Medical University of Lodz, Lodz
  - Central Clinical Hospital of the Ministry of National Defense - Military Institute of Medicine, Warsaw
- Sf. Maria Hospital - University of Medicine and Pharmacy "Carol Davila", Bucharest, Romania
- Saudi Arabia (3):
  - Jazan University, Jizan
  - King Faisal Specialist Hospital and Research Center, Riyadh
  - King Saud University, Riyadh
- Spain (8):
  - Hospital Universitario Cruces - Instituto de investigación sanitaria Biocruces, Barakaldo
  - Hospital Universitario Cruces, Barakaldo
  - Hospital Clinic of Barcelona, Barcelona
  - Hospital Fundación Jiménez Díaz, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario Fundación Jiménez Díaz/Hospital Universitario Rey Juan Carlos, Madrid
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitari Doctor Peset, Valencia
- Farhat Hached Hospital, Sousse, Tunisia
- Turkey (Türkiye) (11):
  - Çukurova University, Adana
  - Ankara Yıldırım Beyazıt University, Ankara
  - Gazi University, Ankara
  - Hacettepe University Faculty of Medicine, Ankara
  - Başakşehir Çam and Sakura City Hospital, Istanbul
  - Cerrahpasa Medical School Istanbul University, Istanbul
  - Marmara University, Research And Education Hospital, Istanbul
  - Dokuz Eylul University School of Medicine, Izmir
  - Manisa Celal Bayar University, Manisa
  - Sakarya University, Sakarya
  - Sivas Cumhuriyet University, Sivas
- I. Horbachevsky Ternopil National Medical University - Ternopil Regional Children's Hospital, Ternopil, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaggiano C, Vitale A, Obici L, Merlini G, Soriano A, Viapiana O, Cattalini M, Maggio MC, Lopalco G, Montin D, Jaber MA, Dagna L, Manna R, Insalaco A, Piga M, La Torre F, Berlengiero V, Gelardi V, Ciarcia L, Emmi G, Ruscitti P, Caso F, Cimaz R, Hernandez-Rodriguez J, Parronchi P, Sicignano LL, Verrecchia E, Iannone F, Sota J, Grosso S, Salvarani C, Frediani B, Giacomelli R, Mencarelli MA, Renieri A, Rigante D, Cantarini L. Clinical Features at Onset and Genetic Characterization of Pediatric and Adult Patients with TNF-alpha Receptor-Associated Periodic Syndrome (TRAPS): A Series of 80 Cases from the AIDA Network. Mediators Inflamm. 2020 Aug 7;2020:8562485. doi: 10.1155/2020/8562485. eCollection 2020. PMID 32831641
- [Background] Vitale A, Sota J, Obici L, Ricco N, Maggio MC, Cattalini M, Ruscitti P, Caso F, Manna R, Viapiana O, Caggiano V, Emmi G, Insalaco A, Montin D, Licciardi F, Soriano A, Dagna L, Salvarani C, Lamacchia V, Hernandez-Rodriguez J, Giacomelli R, Frediani B, Renieri A, Cantarini L. Role of Colchicine Treatment in Tumor Necrosis Factor Receptor Associated Periodic Syndrome (TRAPS): Real-Life Data from the AIDA Network. Mediators Inflamm. 2020 May 27;2020:1936960. doi: 10.1155/2020/1936960. eCollection 2020. PMID 32565720
- [Background] Gaggiano C, Rigante D, Hernandez-Rodriguez J, Vitale A, Tarsia M, Soriano A, Lopalco G, Iannone F, Abdel Jaber M, Giacomelli R, Wiesik-Szewczyk E, Cattalini M, Frassi M, Piga M, Ragab G, Sota J, Zunica F, Floris A, Sabato V, Hegazy MT, Araujo O, Pelegrin L, Fabbiani A, Renieri A, Grosso S, Fabiani C, Frediani B, Cantarini L. Anakinra and canakinumab for patients with R92Q-associated autoinflammatory syndrome: a multicenter observational study from the AIDA Network. Ther Adv Musculoskelet Dis. 2021 Sep 9;13:1759720X211037178. doi: 10.1177/1759720X211037178. eCollection 2021. PMID 34527082
- [Background] Sota J, Rigante D, Cimaz R, Cattalini M, Frassi M, Manna R, Sicignano LL, Verrecchia E, Aragona E, Maggio MC, Lopalco G, Emmi G, Parronchi P, Cauli A, Wiesik-Szewczyk E, Hernandez-Rodriguez J, Gaggiano C, Tarsia M, Mourabi M, Ragab G, Vitale A, Fabiani C, Frediani B, Lamacchia V, Renieri A, Cantarini L; Autoinflammatory Diseases Alliance (AIDA) and the Autoinflammatory Diseases Working Group of the Italian Society of Rheumatology (SIR). Drug survival of anakinra and canakinumab in monogenic autoinflammatory diseases: observational study from the International AIDA Registry. Rheumatology (Oxford). 2021 Dec 1;60(12):5705-5712. doi: 10.1093/rheumatology/keab419. PMID 33961014
- [Background] Sota J, Rigante D, Lopalco G, Emmi G, Gentileschi S, Gaggiano C, Ciarcia L, Berlengiero V, Mourabi M, Ricco N, Barneschi S, Mattioli I, Tosi GM, Frediani B, Tarsia M, di Scala G, Vitale A, Iannone F, Fabiani C, Cantarini L. Clinical profile and evolution of patients with juvenile-onset Behcet's syndrome over a 25-year period: insights from the AIDA network. Intern Emerg Med. 2021 Nov;16(8):2163-2171. doi: 10.1007/s11739-021-02725-9. Epub 2021 Apr 9. PMID 33835406
- [Background] Vitale A, Obici L, Cattalini M, Lopalco G, Merlini G, Ricco N, Soriano A, La Torre F, Verrecchia E, Insalaco A, Dagna L, Jaber MA, Montin D, Emmi G, Ciarcia L, Barneschi S, Parronchi P, Ruscitti P, Maggio MC, Viapiana O, Sota J, Gaggiano C, Giacomelli R, Sicignano LL, Manna R, Renieri A, Lo Rizzo C, Frediani B, Rigante D, Cantarini L. Biotechnological Agents for Patients With Tumor Necrosis Factor Receptor Associated Periodic Syndrome-Therapeutic Outcome and Predictors of Response: Real-Life Data From the AIDA Network. Front Med (Lausanne). 2021 Jul 8;8:668173. doi: 10.3389/fmed.2021.668173. eCollection 2021. PMID 34307404
- [Derived] Tarsia M, Vitale A, Gaggiano C, Sota J, Maselli A, Bellantonio C, Guerriero S, Dammacco R, La Torre F, Ragab G, Hegazy MT, Fonollosa A, Paroli MP, Del Giudice E, Maggio MC, Cattalini M, Fotis L, Conti G, Mauro A, Civino A, Diomeda F, de-la-Torre A, Cifuentes-Gonzalez C, Tharwat S, Hernandez-Rodriguez J, Gomez-Caverzaschi V, Pelegrin L, Babu K, Gupta V, Minoia F, Ruscitti P, Costi S, Breda L, La Bella S, Conforti A, Mazzei MA, Carreno E, Amin RH, Grosso S, Frediani B, Tosi GM, Balistreri A, Cantarini L, Fabiani C. Effectiveness and Safety of Biosimilars in Pediatric Non-infectious Uveitis: Real-Life Data from the International AIDA Network Uveitis Registry. Ophthalmol Ther. 2024 Mar;13(3):761-774. doi: 10.1007/s40123-023-00863-1. Epub 2024 Jan 11. PMID 38206518
- [Derived] Ruscitti P, Sota J, Vitale A, Lopalco G, Iannone F, Morrone M, Giardini HAM, D'Agostin MA, Antonelli IPB, Almaghlouth I, Asfina KN, Khalil N, Sfikakis PP, Laskari K, Tektonidou M, Ciccia F, Iacono D, Riccio F, Ragab G, Hussein MA, Govoni M, Ruffilli F, Direskeneli H, Alibaz-Oner F, Giacomelli R, Navarini L, Bartoloni E, Riccucci I, Martin-Nares E, Torres-Ruiz J, Cipriani P, Di Cola I, Hernandez-Rodriguez J, Gomez-Caverzaschi V, Dagna L, Tomelleri A, Makowska J, Brzezinska O, Iagnocco A, Bellis E, Caggiano V, Gaggiano C, Tarsia M, Mormile I, Emmi G, Sfriso P, Monti S, Erten S, Del Giudice E, Lubrano R, Conti G, Olivieri AN, Lo Gullo A, Tharwat S, Karamanakos A, Gidaro A, Maggio MC, La Torre F, Cardinale F, Ogunjimi B, Maier A, Sebastiani GD, Opris-Belinski D, Frassi M, Viapiana O, Bizzi E, Carubbi F, Fotis L, Tufan A, Kardas RC, Wiesik-Szewczyk E, Jahnz-Rozyk K, Fabiani C, Frediani B, Balistreri A, Rigante D, Cantarini L. The administration of methotrexate in patients with Still's disease, "real-life" findings from AIDA Network Still Disease Registry. Semin Arthritis Rheum. 2023 Oct;62:152244. doi: 10.1016/j.semarthrit.2023.152244. Epub 2023 Jul 21. PMID 37517110
- [Derived] Gaggiano C, Maselli A, Sfikakis PP, Laskari K, Ragab G, Hegazy MT, Laymouna AH, Lopalco G, Almaghlouth IA, Asfina KN, Alahmed O, Giardini Mayrink HA, Parente de Brito Antonelli I, Cattalini M, Piga M, Sota J, Gentileschi S, Maggio MC, Opris-Belinski D, Hatemi G, Insalaco A, Olivieri AN, Tufan A, Karadeniz H, Kardas RC, La Torre F, Cardinale F, Marino A, Guerriero S, Ruscitti P, Tarsia M, Vitale A, Caggiano V, Telesca S, Iannone F, Parretti V, Frassi M, Aragona E, Ciccia F, Wiesik-Szewczyk E, Ionescu R, Sahin A, Akkoc N, Hinojosa-Azaola A, Tharwat S, Hernandez-Rodriguez J, Espinosa G, Conti G, Del Giudice E, Govoni M, Emmi G, Fabiani C, Balistreri A, Frediani B, Rigante D, Cantarini L; AIDA Network. Musculoskeletal manifestations in children with Behcet's syndrome: data from the AIDA Network Behcet's Syndrome Registry. Intern Emerg Med. 2023 Apr;18(3):743-754. doi: 10.1007/s11739-023-03215-w. Epub 2023 Mar 7. PMID 36881285
- [Derived] Gaggiano C, Vitale A, Tufan A, Ragab G, Aragona E, Wiesik-Szewczyk E, Ait-Idir D, Conti G, Iezzi L, Maggio MC, Cattalini M, Torre F, Lopalco G, Verrecchia E, de Paulis A, Sahin A, Insalaco A, Sfikakis PP, Marino A, Frassi M, Ogunjimi B, Opris-Belinski D, Parronchi P, Emmi G, Shahram F, Ciccia F, Piga M, Hernandez-Rodriguez J, Pereira RMR, Alessio M, Naddei R, Olivieri AN, Giudice ED, Sfriso P, Ruscitti P, Gobbi FL, Kucuk H, Sota J, Hussein MA, Malizia G, Jahnz-Rozyk K, Sari-Hamidou R, Romeo M, Ricci F, Cardinale F, Iannone F, Casa FD, Natale MF, Laskari K, Giani T, Franceschini F, Sabato V, Yildirim D, Caggiano V, Hegazy MT, Marzo RD, Kucharczyk A, Khellaf G, Tarsia M, Almaghlouth IA, Laymouna AH, Mastrorilli V, Dotta L, Benacquista L, Grosso S, Crisafulli F, Parretti V, Giordano HF, Mahmoud AAA, Nuzzolese R, Musso M, Chighizola CB, Gentileschi S, Morrone M, Cola ID, Spedicato V, Giardini HAM, Vasi I, Renieri A, Fabbiani A, Mencarelli MA, Frediani B, Balistreri A, Tosi GM, Fabiani C, Lidar M, Rigante D, Cantarini L. The Autoinflammatory Diseases Alliance Registry of monogenic autoinflammatory diseases. Front Med (Lausanne). 2022 Sep 9;9:980679. doi: 10.3389/fmed.2022.980679. eCollection 2022. PMID 36160138
- [Derived] Della Casa F, Vitale A, Cattalini M, La Torre F, Capozio G, Del Giudice E, Maggio MC, Conti G, Alessio M, Ogunjimi B, Ragab G, Emmi G, Aragona E, Giani T, Lopalco G, Parronchi P, Shahram F, Verrecchia E, Ricci F, Cardinale F, Di Noi S, Nuzzolese R, Lubrano R, Patroniti S, Naddei R, Sabato V, Hussein MA, Dotta L, Mastrorilli V, Gentileschi S, Tufan A, Caggiano V, Hegazy MT, Sota J, Almaghlouth IA, Ibrahim A, Wiesik-Szewczyk E, Ozkiziltas B, Grosso S, Frassi M, Tarsia M, Pereira RMR, Taymour M, Gaggiano C, Colella S, Fabiani C, Morrone M, Ruscitti P, Frediani B, Spedicato V, Giardini HAM, Balistreri A, Rigante D, Cantarini L. Development and implementation of the AIDA International Registry for patients with Periodic Fever, Aphthous stomatitis, Pharyngitis, and cervical Adenitis syndrome. Front Pediatr. 2022 Jul 22;10:930305. doi: 10.3389/fped.2022.930305. eCollection 2022. PMID 35935379
- [Derived] Vitale A, Caggiano V, Della Casa F, Hernandez-Rodriguez J, Frassi M, Monti S, Tufan A, Telesca S, Conticini E, Ragab G, Lopalco G, Almaghlouth I, Pereira RMR, Yildirim D, Cattalini M, Marino A, Giani T, La Torre F, Ruscitti P, Aragona E, Wiesik-Szewczyk E, Del Giudice E, Sfikakis PP, Govoni M, Emmi G, Maggio MC, Giacomelli R, Ciccia F, Conti G, Ait-Idir D, Lomater C, Sabato V, Piga M, Sahin A, Opris-Belinski D, Ionescu R, Bartoloni E, Franceschini F, Parronchi P, de Paulis A, Espinosa G, Maier A, Sebastiani GD, Insalaco A, Shahram F, Sfriso P, Minoia F, Alessio M, Makowska J, Hatemi G, Akkoc N, Li Gobbi F, Gidaro A, Olivieri AN, Al-Mayouf SM, Erten S, Gentileschi S, Vasi I, Tarsia M, Mahmoud AAA, Frediani B, Fares Alzahrani M, Laymouna AH, Ricci F, Cardinale F, Jahnz-Rozyk K, Tosi GM, Crisafulli F, Balistreri A, Dagostin MA, Ghanema M, Gaggiano C, Sota J, Di Cola I, Fabiani C, Giardini HAM, Renieri A, Fabbiani A, Carrer A, Bocchia M, Caroni F, Rigante D, Cantarini L. Development and Implementation of the AIDA International Registry for Patients With VEXAS Syndrome. Front Med (Lausanne). 2022 Jul 11;9:926500. doi: 10.3389/fmed.2022.926500. eCollection 2022. PMID 35899212
- [Derived] Vitale A, Della Casa F, Ragab G, Almaghlouth IA, Lopalco G, Pereira RM, Guerriero S, Govoni M, Sfikakis PP, Giacomelli R, Ciccia F, Monti S, Ruscitti P, Piga M, Lomater C, Tufan A, Opris-Belinski D, Emmi G, Hernandez-Rodriguez J, Sahin A, Sebastiani GD, Bartoloni E, Akkoc N, Gunduz OS, Cattalini M, Conti G, Hatemi G, Maier A, Parronchi P, Del Giudice E, Erten S, Insalaco A, Li Gobbi F, Maggio MC, Shahram F, Caggiano V, Hegazy MT, Asfina KN, Morrone M, Prado LL, Dammacco R, Ruffilli F, Arida A, Navarini L, Pantano I, Cavagna L, Conforti A, Cauli A, Marucco EM, Kucuk H, Ionescu R, Mattioli I, Espinosa G, Araujo O, Karkas B, Canofari C, Sota J, Laymouna AH, Bedaiwi AA, Colella S, Giardini HAM, Albano V, Lo Monaco A, Fragoulis GE, Kardas RC, Berlengiero V, Hussein MA, Ricci F, La Torre F, Rigante D, Wiesik-Szewczyk E, Frassi M, Gentileschi S, Tosi GM, Dagostin MA, Mahmoud AAA, Tarsia M, Alessio G, Cimaz R, Giani T, Gaggiano C, Iannone F, Cipriani P, Mourabi M, Spedicato V, Barneschi S, Aragona E, Balistreri A, Frediani B, Fabiani C, Cantarini L; Autoinflammatory Diseases Alliance (AIDA) Network. Development and implementation of the AIDA International Registry for patients with Behcet's disease. Intern Emerg Med. 2022 Oct;17(7):1977-1986. doi: 10.1007/s11739-022-03038-1. Epub 2022 Jul 14. PMID 35831701
- [Derived] Della Casa F, Vitale A, Lopalco G, Ruscitti P, Ciccia F, Emmi G, Cattalini M, Wiesik-Szewczyk E, Maggio MC, Ogunjimi B, Sfikakis PP, Tufan A, Al-Mayouf SM, Del Giudice E, Aragona E, La Torre F, Sota J, Colella S, Di Cola I, Iacono D, Mattioli I, Jahnz-Rozyk K, Joos R, Laskari K, Gaggiano C, Abbruzzese A, Cipriani P, Rozza G, AlSaleem A, Yildirim D, Tarsia M, Ragab G, Ricci F, Cardinale F, Korzeniowska M, Frassi M, Caggiano V, Saad MA, Pereira RM, Berlengiero V, Gentileschi S, Guerriero S, Giani T, Gelardi V, Iannone F, Giardini HAM, Almaghlouth IA, Kardas RC, Ait-Idir D, Frediani B, Balistreri A, Fabiani C, Rigante D, Cantarini L. Development and Implementation of the AIDA International Registry for Patients With Undifferentiated Systemic AutoInflammatory Diseases. Front Med (Lausanne). 2022 Jun 10;9:908501. doi: 10.3389/fmed.2022.908501. eCollection 2022. PMID 35755024
- [Derived] Vitale A, Della Casa F, Lopalco G, Pereira RM, Ruscitti P, Giacomelli R, Ragab G, La Torre F, Bartoloni E, Del Giudice E, Lomater C, Emmi G, Govoni M, Maggio MC, Maier A, Makowska J, Ogunjimi B, Sfikakis PP, Sfriso P, Gaggiano C, Iannone F, Dagostin MA, Di Cola I, Navarini L, Ahmed Mahmoud AA, Cardinale F, Riccucci I, Paroli MP, Marucco EM, Mattioli I, Sota J, Abbruzzese A, Antonelli IPB, Cipriani P, Tufan A, Fabiani C, Ramadan MM, Cattalini M, Kardas RC, Sebastiani GD, Giardini HAM, Hernandez-Rodriguez J, Mastrorilli V, Wiesik-Szewczyk E, Frassi M, Caggiano V, Telesca S, Giordano HF, Guadalupi E, Giani T, Renieri A, Colella S, Cataldi G, Gentile M, Fabbiani A, Al-Maghlouth IA, Frediani B, Balistreri A, Rigante D, Cantarini L. Development and Implementation of the AIDA International Registry for Patients With Still's Disease. Front Med (Lausanne). 2022 Apr 7;9:878797. doi: 10.3389/fmed.2022.878797. eCollection 2022. PMID 35463015
- See also: Website of the AIDA Network — https://aidanetwork.org/en/